CLINICAL TRIAL: NCT01045850
Title: Multicenter, Prospective Cohort of Patient With Coronary Stents Undergoing Non Cardiac Surgery or Invasive Procedures.
Brief Title: Prospective Cohort of Patient With Coronary Stents Undergoing Non Cardiac Surgery
Acronym: RECO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Professor ALBALADEJO Pierre, University Hospital Grenoble
Other Study IDs: DTCIC-09-29; CFAR (Other: Collège Français d'Anesthésie Réanimation)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Cardiovascular Complications; Hemorrhagic Complications
Keywords: coronary stents; non cardiac surgery; cardiovascular complications; hemorrhagic complications; antiplatelet agents; bare metal stent; drug eluting stent; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non cardiac surgery in patients with coronary stents is complicated with cardiovascular and hemorrhagic events associated with perioperative management of antiplatelet agents. Several guidelines have outlined the importance of maintaining antiplatelet agents throughout surgical procedures to prevent cardiovascular complications. On the other hand, interruption of antiplatelet agents is still a usual standard to avoid surgical complications. We investigate the impact of perioperative antiplatelet drugs management on these complications, through a multicenter, prospective cohort (RECO stands for "Registre des patients porteurs d'Endoprothèses Coronaires, Opérés de chirurgie non cardiaque"), including all patients with coronary stents undergoing non cardiac surgery or invasive procedures. The aim of this study is primarily to measure the incidence of cardiovascular (including stent thrombosis) and hemorrhagic complications and to identify pre and postoperative risk factors associated with these complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* patient requiring a non cardiac surgery
* patient with a coronary stent
* patient agree for personal health data collection and analysis

Exclusion Criteria:

* patient less than 18 years
* patient unable to understand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary stents undergoing non cardiac surgery or invasive procedures
Sampling Method: Non-Probability Sample
Enrollment: 1312 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Composite cardiovascular and hemorrhagic postoperative complications | 30 days

SECONDARY OUTCOMES:
Postoperative death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ALBALADEJO, MD, Principal Investigator — University Hospital, Grenoble
Locations (53):
- France (53):
  - HOSPITAL, Aix-en-Provence
  - HOSPITAL, Albi
  - HOSPITAL, Amiens
  - HOSPITAL, Angers
  - HOSPITAL, Avignon
  - HOSPITAL, Beaumont
  - HOSPITAL, Berck
  - HOSPITAL, Besançon
  - HOSPITAL, Bordeaux
  - HOSPITAL, Cabestany
  - HOSPITAL, Castres
  - HOSPITAL, Cavaillon
  - HOSPITAL, Chalon En Champagne
  - HOSPITAL, Chenôve
  - HOSPITAL, Clermont-Ferrand
  - HOSPITAL, Cornebarrieu
  - HOSPITAL, Dracy-le-Fort
  - HOSPITAL, Équeurdreville-Hainneville
  - HOSPITAL, Grenoble
  - HOSPITAL, Hyères
  - HOSPITAL, Istres
  - HOSPITAL, La Roche-sur-Yon
  - HOSPITAL, La Rochelle
  - HOSPITAL, La Seyne-sur-Mer
  - HOSPITAL, Le Mans
  - HOSPITAL, Lyon
  - HOSPITAL, Manosque
  - HOSPITAL, Mantes-la-Jolie
  - HOSPITAL, Marseille
  - HOSPITAL, Maubeuge
  - HOSPITAL, Metz
  - HOSPITAL, Montpellier
  - HOSPITAL, Mulhouse
  - HOSPITAL, Nancy
  - HOSPITAL, Nantes
  - HOSPITAL, Nice
  - HOSPITAL, Niort
  - HOSPITAL, Paris
  - HOSPITAL, Perpignan
  - HOSPITAL, Pierre-Bénite
  - HOSPITAL, Redon
  - HOSPITAL, Rennes
  - HOSPITAL, Romans
  - HOSPITAL, Rouen
  - HOSPITAL, Saint-Denis
  - HOSPITAL, Saint-Dizier
  - HOSPITAL, Saint-Etienne
  - HOSPITAL, Saint-Herblain
  - HOSPITAL, St-Malo
  - HOSPITAL, Toulouse
  - HOSPITAL, Trélazé
  - HOSPITAL, Villeneuve-sur-Lot
  - HOSPITAL, Voiron

REFERENCES:
- [Derived] Albaladejo P, Charbonneau H, Samama CM, Collet JP, Marret E, Piriou V, Genty C, Bosson JL. Bleeding complications in patients with coronary stents during non-cardiac surgery. Thromb Res. 2014 Aug;134(2):268-72. doi: 10.1016/j.thromres.2014.05.015. Epub 2014 May 15. PMID 24913999
- [Derived] Albaladejo P, Marret E, Samama CM, Collet JP, Abhay K, Loutrel O, Charbonneau H, Jaber S, Thoret S, Bosson JL, Piriou V. Non-cardiac surgery in patients with coronary stents: the RECO study. Heart. 2011 Oct;97(19):1566-72. doi: 10.1136/hrt.2011.224519. Epub 2011 Jul 26. PMID 21791513